CLINICAL TRIAL: NCT02113059
Title: "Involvement of Platelets and Platelet Derived Growth Factors in Postoperative Liver Regeneration, Liver Dysfunktion and Morbidity in Patients Undergoing Hepatectomy"
Brief Title: Platelets in Liver Regeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Patrick Starlinger, MD, PhD, Medical University of Vienna
Other Study IDs: PS-AS-TG-CB
Record Dates: First submitted 2014-04-06; First posted 2014-04-14 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Liver Regeneration
Keywords: Liver regeneration; liver dysfunction; platelets; plasma; serum; platelet activation; morbidity; mortality; Growth factors; Postoperative clinical outcome
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, platelet and tissue preparation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver resection: Patients undergoing a hemihepatectomy.

SUMMARY:
The most relevant factor predicting morbidity and mortality after liver resections is the ability of the remnant liver to regenerate. The investigators recently demonstrated that serotonin and thrombospondin-1, two growth factors abundantly stored in platelets, seem to play a critical role in liver regeneration of patients after liver resection. The investigators now aim to gain more precise insight concerning the relevance of platelets and platelet derived growth factors in liver regeneration in humans. The investigators will focus on specific alpha-granula release as a key regulator of postoperative LR. Using peri- and intraoperative blood and tissue samples, platelet adhesion, granula release and induction of gene expression known to be involved in liver regeneration form experimental studies will be analyzed. This study should allow the investigators to verify observations from preclinical models and evaluate their relevance in the human setting. Furthermore, this might enable the investigators to identify new therapeutic targets.

DETAILED DESCRIPTION:
The investigators could previously show that platelet derived growth factors like TSP-1 and 5-HT are of relevance in human liver regeneration. In this project the investigators aim to elucidate how platelets specifically release their granules. Indeed, while dense granules stored 5-HT induces proliferation of hepatocytes, alpha-granules stored TSP-1 reduces their proliferative potential. More importantly, various pro-proliferative growth factors as VEGF are also stored in alpha-granules. Therefore, a systemic reduction in platelet counts would reduce both, pro and anti-proliferative factors. A highly regulated granula release has been postulated to allow platelets to exert specific functions. In 2008, Italiano et al. presented convincing in vitro evidence that platelets store molecules in separate granules, which they are able to specifically release upon platelet activation. Furthermore, results by other groups support this finding.

It is the aim of this project to characterize platelet activation in patients with liver resection and determine if specific platelet activation profiles correlate with clinical outcome.

Project plan

Included patients:

A total of 40 patients undergoing hemihepatectomy will be included. Patients will be closely monitored perioperatively. Plasma, serum, platelet and tissue preparation will be performed as outlined below.

Hypothesis No. 1:

Circulating platelet activation markers increase after liver resection.

To confirm the investigators initial observation of specific granula release, platelet activation will be monitored during liver regeneration. In particular, the investigators will evaluate platelet activation markers during the perioperative period. In a descriptive manner, the investigators will identify perioperative fluctuations of platelet activation as a reflection of physiologic processes during liver regeneration. This should enable the investigators to elucidate the occurrence of platelet activation in the human setting, as it has been described in murine models. More importantly, the investigators analyses could identify potential treatment targets in patients with insufficient hepatic regeneration.

Hypothesis No. 2:

Intra platelet granula contents decrease after liver resection.

Bioactive molecules stored in platelet alpha granules (intra platelet - IP), will be evaluated during the perioperative period. As during serum preparation all platelets degranulate, IP levels of granula contents will be calculated by subtraction of plasma from serum growth factor values. Furthermore to confirm these calculated values, platelet extracts will be generated and comparatively analyzed for IP growth factor levels. The investigators will further be able to identify perioperative fluctuations of IP growth factors as a reflection of specific intrahepatic release during liver regeneration, by comparing blood samples prior and one day after liver resection.

Hypothesis No. 3:

Platelets are locally enriched and activated at the site of liver regeneration.

During the process of a classical hemihepatectomy, the portal vein of the tumor containing liver lobe is initially ligated before mobilization and dissection of the liver. The increase of portal pressure within the remaining liver after partial hepatectomy is believed to be the major inducer of liver regeneration. (37-40) To evaluate if platelets play a critical role during the process of initiation of liver regeneration, tissue specimens will be collected prior to portal vein ligation and one hour after portal vein ligation (at the time of initiation of liver regeneration)(study design is illustrated in figure 3). Liver specimens will then be comparatively analyzed for platelet adhesion and protein as well as mRNA expression.

To further evaluate the relevance of platelets in the tightly regulated process of liver regeneration, blood will be collected 1 hour after portal vein ligation. In particular, blood will be drawn from the portal vein (prior to the liver) and from a liver vein (after the liver). From these samples platelets will be isolated and the degree of activation will be evaluated (details see below). Furthermore, the content of IP growth factors and platelet extracts will be analyzed to reflect their intrahepatic release.

Hypothesis No. 4:

Perioperative platelet activation has an impact on postoperative outcome

The predictive potential of platelet activation markers and IP growth factors to identify patients with poor postoperative clinical outcome will be analyzed. As outcome parameters postoperative LD, morbidity or mortality will be evaluated. These analyses might identify markers to select patients that should not undergo hepatectomy but be better served with alternative treatments. Furthermore, potential treatment targets in patients with insufficient hepatic regeneration could be identified.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective hemihepatectomy

Exclusion Criteria:

* peroperative portal vein thrombosis
* age > 85

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients undergoing elective hemihepatectomy.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Validation of the role of platelets in the process of early liver regeneration in humans | 2 years
  Preclinical studies have identified multiple platelet associated candidate molecules in the highly regulated process of liver regeneration. Using a complex peri and intraoperative sampling schedule, we will try to validate the relevance of these molecules in the human setting.

SECONDARY OUTCOMES:
Postoperative liver dysfunction | 2 years
  Association of peri and intraoperative blood and tissue parameters associated with postoperative liver dysfunction
Postoperative morbidity | 2 years
  Association of peri and intraoperative blood and tissue parameters associated with postoperative morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Starlinger, MD, PhD, Principal Investigator — Medical University Vienna; Alice Assinger, PhD, Principal Investigator — Medical University Vienna
Locations (2):
- Austria (2):
  - Rudolfstiftung, Vienna
  - Medical University Vienna, Vienna